CLINICAL TRIAL: NCT01111136
Title: Effect of Psychological Stress Intervention for Patients With Chronic Urticaria
Brief Title: Stress Intervention for Chronic Urticaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: John W. Tole, D.O., University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2010-0052
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Urticaria
Keywords: Urticaria; Hives; Stress
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stress intervention (Experimental): Stress intervention.
  Interventions: Behavioral: Stress intervention

INTERVENTIONS:
Behavioral: Stress intervention — To evaluate psychological stress, participants will complete the Perceived Stress Scale, Beck Depression Inventory-Fast Screen, Anxiety Sensitivity Index-III, Posttraumatic Stress Diagnostic Scale and the Depression Anxiety Stress Scales; to evaluate cognitive and behavioral aspects of emotional avoidance, participants will complete the Emotional Avoidance Questionnaire as well as the Acceptance and Action Questionnaire, Difficulties in Emotion Regulation Scale, Illness Attitudes Scale and the Five Facet Mindfulness Questionnaire; and to evaluate quality of life in regards to his/her skin condition, participants will complete the Dermatology Life Quality Index questionnaire.

SUMMARY:
Stress and chronic urticaria has been linked. The purpose of the study is to evaluate a patients chronic urticaria and stress levels before and after he/she goes through six sessions designed to help that participant manage his/her stress.

DETAILED DESCRIPTION:
The purpose of this single-arm, interventional pilot study is to evaluate the effect of psychological stress intervention for patients with chronic urticaria, as many of these patients report heightened levels of stress before and/or after the onset of the urticaria. Participants will meet individually with a University of Mississippi Medical Center psychiatry resident for one hour once a week for six consecutive weeks to be educated on psychological stress intervention techniques. There is no control group for this pilot study. All participants will complete a packet of psychological and dermatological questionnaires before the first session with the psychiatry resident and one week after the final session. All participants will record daily 1) their urticaria symptoms and 2) the type and number of medications taken for his/her chronic hives. If psychological stress intervention proves to be effective, then this therapeutic modality would benefit patients with chronic urticaria, while avoiding addition and/or continuation of medications that may have significant adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-64 years old who have had hives for longer than 6 weeks.
* Hives persist despite medical therapy.
* Minimum Urticaria Activity Score of 2 (one point from each of the two categories: number of hives and severity of pruritus).

Exclusion Criteria:

* Urticaria secondary to vasculitis.
* Urticaria as part of an anaphylactic response.
* Use of Omalizumab within 3 months preceding enrollment period.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Urticaria Activity Score | 7 weeks
  Measures the daily level of skin itching and the number of hives as the study progresses.

SECONDARY OUTCOMES:
Level of stress. | 7 weeks
  A set of questionnaires done before the first session and after the sixth/final session will be done to compare level of stress.

CONTACTS AND LOCATIONS:
Overall Officials: John W. Tole, D.O., Principal Investigator — University of Mississippi Medical Center; Gailen D. Marshall, MD, PhD, Study Director — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Powell RJ, Du Toit GL, Siddique N, Leech SC, Dixon TA, Clark AT, Mirakian R, Walker SM, Huber PA, Nasser SM; British Society for Allergy and Clinical Immunology (BSACI). BSACI guidelines for the management of chronic urticaria and angio-oedema. Clin Exp Allergy. 2007 May;37(5):631-50. doi: 10.1111/j.1365-2222.2007.02678.x. PMID 17456211
- [Background] Sperber J, Shaw J, Bruce S. Psychological components and the role of adjunct interventions in chronic idiopathic urticaria. Psychother Psychosom. 1989;51(3):135-41. doi: 10.1159/000288147. PMID 2636418
- [Background] Papadopoulou N, Kalogeromitros D, Staurianeas NG, Tiblalexi D, Theoharides TC. Corticotropin-releasing hormone receptor-1 and histidine decarboxylase expression in chronic urticaria. J Invest Dermatol. 2005 Nov;125(5):952-5. doi: 10.1111/j.0022-202X.2005.23913.x. PMID 16297195
- [Background] Yang HY, Sun CC, Wu YC, Wang JD. Stress, insomnia, and chronic idiopathic urticaria--a case-control study. J Formos Med Assoc. 2005 Apr;104(4):254-63. PMID 15909063
- [Background] Ozkan M, Oflaz SB, Kocaman N, Ozseker F, Gelincik A, Buyukozturk S, Ozkan S, Colakoglu B. Psychiatric morbidity and quality of life in patients with chronic idiopathic urticaria. Ann Allergy Asthma Immunol. 2007 Jul;99(1):29-33. doi: 10.1016/S1081-1206(10)60617-5. PMID 17650826
- [Background] Silvares MR, Coelho KI, Dalben I, Lastoria JC, Abbade LP. Sociodemographic and clinical characteristics, causal factors and evolution of a group of patients with chronic urticaria-angioedema. Sao Paulo Med J. 2007 Sep 6;125(5):281-5. doi: 10.1590/s1516-31802007000500006. PMID 18094895
- [Background] Berrino AM, Voltolini S, Fiaschi D, Pellegrini S, Bignardi D, Minale P, Troise C, Maura E. Chronic urticaria: importance of a medical-psychological approach. Eur Ann Allergy Clin Immunol. 2006 May;38(5):149-52. PMID 17058846
- [Background] Annesi-Maesano I, Beyer A, Marmouz F, Mathelier-Fusade P, Vervloet D, Bauchau V. Do patients with skin allergies have higher levels of anxiety than patients with allergic respiratory diseases? Results of a large-scale cross-sectional study in a French population. Br J Dermatol. 2006 Jun;154(6):1128-36. doi: 10.1111/j.1365-2133.2006.07186.x. PMID 16704645